CLINICAL TRIAL: NCT00336193
Title: University of Colorado Health Sciences Center: Competency Training, Staff Performance, & Family Outcomes
Brief Title: Competency Training, Staff Performance, & Family Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Ruth O'Brien, University of Colorado Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCIPC-4537
Record Dates: First submitted 2006-06-10; First posted 2006-06-13 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Child Abuse
Keywords: home visitation; family outcomes; competency training

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home visitation (Experimental): In the intervention condition, nurse home visitors receive enhanced training to improve delivery of parenting interventions to mothers
  Interventions: Behavioral: Home visitation

INTERVENTIONS:
Behavioral: Home visitation — Home visitation to improve maternal health and well-being and parenting practices

SUMMARY:
This proposal examines the impact of an augmented competency based approach to training of home visitors and supervisors for delivery of the Nurse Family Partnership (NFP) on staff performance, fidelity to the program model, and family outcomes relative to child maltreatment and early behaviors associated with youth violence. The central premise underlying the proposed study is that the augmented competency based curriculum and clinical consultation to supervisors will improve nurses' knowledge and skills in working with families, which in turn, will lead to greater fidelity to the home visit guidelines (i.e., quality implementation), which in turn, will result in better maternal and child health outcomes.

DETAILED DESCRIPTION:
A two group experimental design will be used to examine the impact of an augmented competency-based curriculum for NFP home visitors and supervisors coupled with structured clinical consultation by NFP National Office professional development staff, as compared against the standard curriculum currently used, on quality of program implementation and family outcomes.

ELIGIBILITY:
Inclusion Criteria:

* First time mothers (enrolled during pregnancy) and their children

Exclusion Criteria:

* See above. No other exclusion criteria will be used.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1075 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Assessment of children's home environment | 12 and 24 months
Children's emergency room visits/hospitalizations | 6, 12, 18, and 24 months
Children's adjustment and behavior | 21-22 months
Children's language development at 21 months | 21 months
Referrals to child protective services 6, 12, 18, and 24 months | 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A O'Brien, RN PhD, Principal Investigator — University of Colorado Denver Health Sciences Center
Locations (1):
- University of Colorado Denver Health Sciences Center, Denver, Colorado, United States